CLINICAL TRIAL: NCT00837473
Title: A Prospective Pilot Study on the Performance of The Plexur P™ Bone Void Filler
Brief Title: Study Performance of The Plexur P™ Bone Void Filler Device in Patients Undergoing Iliac Crest Harvesting Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Osteotech, Inc (Industry)
Responsible Party: Sponsor
Organization: Medtronic Spinal and Biologics (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Trial #3206
Record Dates: First submitted 2009-02-04; First posted 2009-02-05 (Estimated); Results first posted 2018-04-30 (Actual); Last update posted 2018-04-30 (Actual); Status verified 2012-09

CONDITIONS: Iliac Crest Harvesting Procedure-Bone Void Filler
Keywords: Bone Void Filler; Iliac Crest Bone Void Filler; Back Surgery and Autograft Bone; Autograft Bone; Allograft Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Plexur-P Bone Void Filler (Other): Single arm. Open Label.
  Interventions: Device: Plexur-P used as a Bone Void Filler in Iliac Crest Harvesting Procedures

INTERVENTIONS:
Device: Plexur-P used as a Bone Void Filler in Iliac Crest Harvesting Procedures — Plexur-P used as a Bone Void Filler in Iliac Crest Harvesting Procedures

SUMMARY:
The purpose of this study is to determine if Plexur P grows bone in the iliac crest (where bone was removed or "harvested") for the back surgery.

The study will be focusing on patients who require back surgery. Often additional bone is required from the hip of the patient (iliac crest). When bone removed from the hip, a "void" is often created. This "void" will be filled in with Osteotech's Plexur P product.

DETAILED DESCRIPTION:
This prospective trial is designed to evaluate the ability of the Plexur P device (bone void filler) to reconstitute the iliac crest in patients requiring iliac crest bone harvesting procedures at one single study site.

Plexur P Bone Void Filler is:

* A biocomposite of mineralized cortical allograft bone fibers and polylactide-co-glycolide co-polymer.
* Designed to fill bony voids or gaps of the skeletal system that are not intrinsic to the stability of the bony structure.
* Porosity is introduced into the Plexur P Biocomposites to create a cancellous-like structure that provides a scaffold for bone growth.

In addition:

* Patients will be screened for study eligibility based on the need for iliac crest bone harvesting.
* Fifteen (15) eligible patients will be enrolled and will have an iliac crest harvesting defect backfilled with Plexur P to repair the iliac crest defect.
* As a part of routine follow up care, patient related outcomes including measurements of pain severity and pain relief will be determined using patient (IRB approved) questionnaires.
* Radiographic analysis will also be used to determine amount of bony ingrowth of the Plexur P device.

ELIGIBILITY:
Inclusion Criteria:

* The patient is at least 18 yrs old.
* The patient requires an iliac crest harvesting procedure.
* The patient has signed an Informed Consent, approved by the IRB.

Exclusion Criteria:

* Patient is less than 18 years old.
* Patient presents with a bony void or gap in an area other than the iliac crest and/or has an infection present at the (operative) site.
* Insulin dependent diabetics and/or in the opinion of the investigator, has poorly controlled non-insulin dependent diabetes.
* The patient is a smoker.
* The patient is mentally compromised (e.g., currently being treated from a psychiatric disorder, senile dementia, Alzheimer's disease, etc.) and/or in the opinion of the investigator, is not likely to complete follow up visits;
* The patient has a bleeding disorder of any etiology, severe vascular or neurological disease;
* The patient has hypercalcemia and/or severe degenerative bone disease;
* The patient has a history of long term steroid use;
* The patient requires immunosuppressive therapy;
* The patient has a history of drug or alcohol abuse that may interfere with his/her ability to provide written informed consent;
* The patient is pregnant at the time of study entry or may likely become pregnant during the course of study participation;
* The subject has an implanted device, which is incompatible with the use of imaging equipment;
* The patient has an allergy to one of the components of the investigational device;
* The patient has renal insufficiency;
* The patient has a terminal illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-01; Primary Completion 2011-03 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oheneba Boachie-Adijei, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Plexur-P Bone Void Filler
Started | 15
Completed | 12
Not Completed | 3
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Plexur-P Bone Void Filler
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.13 (9.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Reconstitution of Bone Growth in the Iliac Crest Bone Void Determined by an Independent Radiologist
Description: Reconstitution of bone growth was determined by an independent radiologist based on bony ingrowth and absence of a gap according to the following criteria:
  * Absent: limited or no bone mineralization visualized at the defect site; extensive areas of radiolucency.
  * Mild: identifiable bone mineralization and coalescence of the bone graft mass of < 50% of the defect site.
  * Moderate: identifiable bone mineralization and coalescence of the bone graft mass over > 50% of the defect site; some remaining unmineralized areas of radiolucency; limited evidence of partial bone remodeling and trabeculation.
  * Extensive: > 75% of bone mineralization over the defect site showing a contiguous and completely coalesced bone graft mass with confluent trabecular pattern.
Time Frame: 6 wks, 3 mths, 6 mths 12 mths, and 24 mths
Population: The primary analysis dataset included all study subjects with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Plexur-P Bone Void Filler
Number analyzed (Participants) | 15
Participants
  Reconstitution at 6 weeks: Absent | 11
  Reconstitution at 6 weeks: Mild | 4
  Reconstitution at 6 weeks: Moderate | 0
  Reconstitution at 6 weeks: Extensive | 0
  Reconstitution at 3 months: number analyzed (Participants) | 5
  Reconstitution at 3 months: Absent | 3
  Reconstitution at 3 months: Mild | 1
  Reconstitution at 3 months: Moderate | 1
  Reconstitution at 3 months: Extensive | 0
  Reconstitution at 6 months: number analyzed (Participants) | 12
  Reconstitution at 6 months: Absent | 0
  Reconstitution at 6 months: Mild | 10
  Reconstitution at 6 months: Moderate | 2
  Reconstitution at 6 months: Extensive | 0
  Reconstitution at 12 months: number analyzed (Participants) | 13
  Reconstitution at 12 months: Absent | 0
  Reconstitution at 12 months: Mild | 6
  Reconstitution at 12 months: Moderate | 6
  Reconstitution at 12 months: Extensive | 1
  Reconstitution at 24 months: number analyzed (Participants) | 12
  Reconstitution at 24 months: Absent | 0
  Reconstitution at 24 months: Mild | 1
  Reconstitution at 24 months: Moderate | 9
  Reconstitution at 24 months: Extensive | 2

2. Secondary Outcome: General Health Status
Description: The general health status was assessed by Medical Outcomes Study 36-Item Short Form Health Survey (SF-36v2). The SF-36v2 questionnaire contains 36 questions pertaining to eight subscales of health status. These eight subscales can be summarized as relating to either physical health or mental health. The physical component summary (PCS) is based primarily on the physical functioning, role-physical, bodily pain, and general health scales of the SF-36v2 survey. The mental component summary (MCS) encompasses vitality, social functioning, role-emotional, and mental health scales. The score for PCS and MCS is between 0 and 100, with higher scores denoting better quality of life.
Time Frame: Baseline, 6 wks, 3 mths, 6 mths, 12 mths, and 24 mths
Population: The primary analysis dataset included all study subjects with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Plexur-P Bone Void Filler
Number analyzed (Participants) | 15
units on a scale
  SF-36 PCS score at baseline: number analyzed (Participants) | 10
  SF-36 PCS score at baseline | 35.36 (8.67)
  SF-36 PCS score at 6 weeks: number analyzed (Participants) | 9
  SF-36 PCS score at 6 weeks | 29.41 (8.51)
  SF-36 PCS score at 3 months: number analyzed (Participants) | 3
  SF-36 PCS score at 3 months | 35.68 (10.36)
  SF-36 PCS score at 6 months: number analyzed (Participants) | 9
  SF-36 PCS score at 6 months | 41.68 (10.77)
  SF-36 PCS score at 12 months: number analyzed (Participants) | 11
  SF-36 PCS score at 12 months | 41.23 (12.25)
  SF-36 PCS score at 24 months: number analyzed (Participants) | 9
  SF-36 PCS score at 24 months | 37.43 (14.90)
  SF-36 MCS score at baseline: number analyzed (Participants) | 10
  SF-36 MCS score at baseline | 43.86 (12.74)
  SF-36 MCS score at 6 weeks: number analyzed (Participants) | 9
  SF-36 MCS score at 6 weeks | 45.91 (14.38)
  SF-36 MCS score at 3 months: number analyzed (Participants) | 3
  SF-36 MCS score at 3 months | 54.50 (9.98)
  SF-36 MCS score at 6 months: number analyzed (Participants) | 9
  SF-36 MCS score at 6 months | 50.36 (16.24)
  SF-36 MCS score at 12 months: number analyzed (Participants) | 11
  SF-36 MCS score at 12 months | 49.69 (12.72)
  SF-36 MCS score at 24 months: number analyzed (Participants) | 9
  SF-36 MCS score at 24 months | 44.87 (11.35)

3. Secondary Outcome: Oswestry Disability Index
Description: The Oswestry Disability Index (ODI) is an internationally validated questionnaire consisting of ten sets of statements which focus on pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sex life, social life, and ability to travel. ODI scores are in a range of 0 to 100, with a lower score indicating less pain and disability and higher scores indicating more pain and disability.
Time Frame: Baseline, 6 wks, 3 mths, 6 mths, 12 mths, and 24 mths
Population: The primary analysis dataset included all study subjects with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Plexur-P Bone Void Filler
Number analyzed (Participants) | 15
units on a scale
  ODI at baseline: number analyzed (Participants) | 11
  ODI at baseline | 54.28 (17.88)
  ODI at 6 wks: number analyzed (Participants) | 12
  ODI at 6 wks | 70.19 (15.95)
  ODI at 3 months: number analyzed (Participants) | 3
  ODI at 3 months | 56.44 (20.26)
  ODI at 6 months: number analyzed (Participants) | 11
  ODI at 6 months | 44.86 (16.71)
  ODI at 12 months: number analyzed (Participants) | 11
  ODI at 12 months | 41.92 (20.03)
  ODI at 24 months: number analyzed (Participants) | 10
  ODI at 24 months | 50.80 (19.94)

4. Secondary Outcome: Pain Status Assessed by Visual Analog Scale (VAS)
Description: The visual analog scale (VAS) was used for assessing pain status in the body locations of back/neck, left leg/arm, and right arm/leg. Subjects were asked to rate their perception of pain in VAS, generated by the Osteotech Clinical Department. The scale from 1 to 5 represented the pain levels at none, mild, average, severe, and extreme.
Time Frame: Baseline, 6 wks, 3 mths, 6 mths, 12 mths, and 24 mths
Population: The primary analysis dataset included all study subjects with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Plexur-P Bone Void Filler
Number analyzed (Participants) | 15
units on a scale
  Back/neck pain at baseline: number analyzed (Participants) | 11
  Back/neck pain at baseline | 3.5 (1.4)
  Back/neck pain at 6 weeks: number analyzed (Participants) | 12
  Back/neck pain at 6 weeks | 2.6 (1.2)
  Back/neck pain at 3 months: number analyzed (Participants) | 3
  Back/neck pain at 3 months | 2.3 (1.5)
  Back/neck pain at 6 months: number analyzed (Participants) | 10
  Back/neck pain at 6 months | 2.4 (1.1)
  Back/neck pain at 12 months: number analyzed (Participants) | 10
  Back/neck pain at 12 months | 2.1 (1.0)
  Back/neck pain at 24 months: number analyzed (Participants) | 9
  Back/neck pain at 24 months | 2.8 (1.5)
  Left leg/arm pain at baseline: number analyzed (Participants) | 9
  Left leg/arm pain at baseline | 2.0 (1.2)
  Left leg/arm pain at 6 weeks: number analyzed (Participants) | 12
  Left leg/arm pain at 6 weeks | 2.1 (1.2)
  Left leg/arm pain at 3 months: number analyzed (Participants) | 3
  Left leg/arm pain at 3 months | 1.7 (0.6)
  Left leg/arm pain at 6 months: number analyzed (Participants) | 10
  Left leg/arm pain at 6 months | 1.7 (0.8)
  Left leg/arm pain at 12 months: number analyzed (Participants) | 10
  Left leg/arm pain at 12 months | 1.9 (1.4)
  Left leg/arm pain at 24 months: number analyzed (Participants) | 7
  Left leg/arm pain at 24 months | 2.0 (1.4)
  Right leg/arm pain at baseline: number analyzed (Participants) | 9
  Right leg/arm pain at baseline | 2.0 (1.1)
  Right leg/arm pain at 6 weeks: number analyzed (Participants) | 12
  Right leg/arm pain at 6 weeks | 1.9 (0.9)
  Right leg/arm pain at 3 months: number analyzed (Participants) | 3
  Right leg/arm pain at 3 months | 1.7 (1.2)
  Right leg/arm pain at 6 months: number analyzed (Participants) | 10
  Right leg/arm pain at 6 months | 1.6 (0.8)
  Right leg/arm pain at 12 months: number analyzed (Participants) | 10
  Right leg/arm pain at 12 months | 1.8 (1.5)
  Right leg/arm pain at 24 months: number analyzed (Participants) | 9
  Right leg/arm pain at 24 months | 2.1 (1.3)

5. Secondary Outcome: Surgical Related Outcome--locations of Iliac Crest Bone Harvest
Time Frame: During the time of operation, a range of 2.5-8.5 hrs
Measure: Count of Participants; unit: Participants
Arm/Group | Plexur-P Bone Void Filler
Number analyzed (Participants) | 15
Participants
  Left side | 8
  Right side | 7

6. Secondary Outcome: Surgical outcome-the Amount of Cancellous Bone Harvested
Time Frame: During the time of operation, a range of 2.5-8.5 hrs
Measure: Mean (Standard Deviation); unit: cc
Arm/Group | Plexur-P Bone Void Filler
Number analyzed (Participants) | 15
cc | 14.6 (5.4)

7. Secondary Outcome: Surgical Outcome--operative Time
Time Frame: The time of operation, a range of 2.5-8.5 hrs
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Plexur-P Bone Void Filler
Number analyzed (Participants) | 15
min | 310.0 (97.2)

8. Secondary Outcome: Surgical Outcome--blood Loss
Time Frame: During the time of operation, a range of 2.5-8.5 hrs
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Plexur-P Bone Void Filler
Number analyzed (Participants) | 15
ml | 1786.7 (1128.8)

9. Secondary Outcome: Surgical Outcome--length of Hospital Stay
Time Frame: From admission to discharge, a range of 2 to 20 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Plexur-P Bone Void Filler
Number analyzed (Participants) | 15
days | 10.7 (4.6)

10. Secondary Outcome: Surgical Outcome- the Amount of Plexur™ P Product Utilized for Filling Void
Time Frame: During the time of operation, a range of 2.5-8.5 hrs
Measure: Mean (Standard Deviation); unit: cc
Arm/Group | Plexur-P Bone Void Filler
Number analyzed (Participants) | 15
cc | 24.7 (5.6)

ADVERSE EVENTS:
Time Frame: Overall study period, up to 24 months
Description: All adverse events that observed by the investigator or reported spontaneously by the study participants were recorded on the Clinical Complication/Adverse Event Form by the investigator.
Arm/Group | Plexur-P Bone Void Filler
Serious Adverse Events (participants affected / at risk) | 12/15
Other Adverse Events (participants affected / at risk) | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Plexur-P Bone Void Filler (N=15)
Other (Endocrine disorders) | 1 (1)
Other (General disorders) | 1 (1)
Infection other (Infections and infestations) | 1 (1)
Other (Infections and infestations) | 1 (1)
Other (Injury, poisoning and procedural complications) | 5 (6)
Other (Metabolism and nutrition disorders) | 1 (1)
Other (Musculoskeletal and connective tissue disorders) | 1 (1)
Other (Nervous system disorders) | 1 (1)
Other (Product Issues) | 3 (4)
Other (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Other (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Plexur-P Bone Void Filler (N=15)
Other (Cardiac disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 3 (3)
Edema (General disorders) | 2 (2)
Other (General disorders) | 1 (1)
Infection, other (Infections and infestations) | 2 (2)
Infection, operative site (Infections and infestations) | 1 (1)
Other (Infections and infestations) | 2 (2)
Other (Injury, poisoning and procedural complications) | 1 (1)
Other (Investigations) | 3 (3)
Other (Metabolism and nutrition disorders) | 1 (1)
Other (Musculoskeletal and connective tissue disorders) | 1 (1)
Other (Nervous system disorders) | 2 (2)
Urine Retention (Renal and urinary disorders) | 1 (1)
Other (Respiratory, thoracic and mediastinal disorders) | 9 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No